CLINICAL TRIAL: NCT03549299
Title: An Interventional, Open-label, Multicenter Phase I/IIa Clinical Trial to Investigate the Safety and Efficacy of Ascending Doses of Allogeneic ABCB5-positive Limbal Stem Cells (LSC2) for the Treatment of Limbal Stem Cell Deficiency (LSCD)
Brief Title: Allogeneic ABCB5-positive Limbal Stem Cells for Treatment of LSCD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Ticeba GmbH (Industry); Granzer Regulatory Consulting & Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSC2-II-01
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: limbal stem cell deficiency; ABCB5; Limbal stem cells; LSCs; LSC; allogeneic; tissue engineered product; phase I/IIa
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Intervention Model Description: Patients will be treated in up to four ascending dose groups. After the first treated patient of the first dose group (Group A) was followed for 2 weeks, a safety and tolerability assessment of the applied IMP dose will be conducted by an internal committee. The same approach applies to the second subject.
  Dose escalation and recruitment of additional patients into the second dose group (Group B) will depend on the safety and tolerability of the IMP in Group A. A safety and tolerability assessment will be conducted after the last treated patient of the first dose group (Group A) was followed for 12 weeks.
  The same approach applies to Group C and D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LSC2; 7.5 x 10^4 cells (Experimental): Single dose of LSC2, 7.5 x 10^4 cells per patient
  Interventions: Biological: LSC2
- LSC2; 3.0 x 10^5 cells (Experimental): Single dose of LSC2, 3.0 x 10^5 cells per patient
  Interventions: Biological: LSC2
- LSC2; 8.0 x 10^5 cells (Experimental): Single dose of LSC2, 8.0 x 10^5 cells per patient
  Interventions: Biological: LSC2
- LSC2; 1.2 x 10^6 cells (Experimental): Single dose of LSC2, 1.2 x 10^6 cells per patient
  Interventions: Biological: LSC2

INTERVENTIONS:
Biological: LSC2 — Topical application of IMP on target eye
  Other Names: Suspension of ABCB5-positive limbal stem cells in pre-filled syringe

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring neovascularization and epithelial defects) of up to four doses of the investigational medicinal product (IMP) LSC2 topically administered on the target eye of patients with LSCD. Further, safety of the IMP during and after application will be investigated (by monitoring adverse events [AEs]).

DETAILED DESCRIPTION:
This is an interventional, open-label, phase I/IIa clinical trial to investigate the efficacy and safety of up to four doses of the IMP topically administered on the target eye of patients with LSCD. Patients will be treated in up to four ascending dose groups.

The allogeneic investigational product LSC2 contains ABCB5-positive limbal stem cells (from corneal rims of cadaveric donors, expanded ex vivo, isolated and stored in a donor cell bank).

The IMP will be applied on the target eye. Prior to application, the conjunctival pannus will be removed under general or local anesthesia.

Patients will be followed up for efficacy for 1 year. Efficacy of the IMP will be monitored by assessing neovascularization and epithelial defects.

To assess long-term safety of LSC2 one follow-up visit at Month 24 post IMP application is included.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 85 years
2. Patients with secondary bilateral or unilateral LSCD (injury that caused LSCD at least 6 months prior to inclusion)
3. Neovascularization: Vessel penetration of at least 2 quadrants, with central cornea involved
4. Patients understand the nature of the procedure and are providing written informed consent prior to any clinical trial procedure
5. Women of childbearing potential must have a negative blood pregnancy test at Visit 1
6. Women of childbearing potential must be willing to use highly effective contraceptive methods during the course of the clinical trial

Exclusion Criteria:

1. Compromised eyelid mobility and/or symblepharon; patient can be re-screened after appropriate treatment
2. Presence of eyelid malposition; patient can be re-screened after appropriate treatment
3. Active local ocular or systemic infection and/or inflammation. Patient can be re-screened after infection and/or inflammation is resolved.
4. Tumor diseases or history of tumor disease
5. Active ocular neoplastic disease (exclusion will be based on investigator's assessment)
6. Corneal erosion or ulcer is bigger than 4 mm2; corresponding to less than 95% of continuous corneal epithelium. Patient can be re-screened after erosion or ulcer is resolved (≤ 4 mm2).
7. Positive for human immunodeficiency virus (HIV) 1 and/or 2 (diagnosed by serologic testing)
8. Clinically significant or unstable concurrent disease or other clinical contraindications to stem cell transplantation
9. History of glaucoma
10. Contraindications to trial related procedures/substances including

    1. The surgical procedure (e.g. removing of the conjunctival pannus)
    2. Contact lens complications due to contact lens use in the proposed trial (based on the Efron Grading scale for standard clinical reference for contact lens complications)
    3. Tear secretion deficiency determined by Schirmer's test
    4. Allergy, sensitivity or intolerance to components/excipients of the IMP/ per protocol pre-planned concomitant medications
    5. Conjunctival scarring with fornix shortening
    6. General anesthesia (in case general anesthesia is required) or local anesthesia
    7. Immunosuppression (being mandatory concomitant therapy)
11. Intraocular pressure (IOP) of ≥30 mm Hg
12. History or clinical signs of stroke or transient ischemic attacks
13. Active or suspected ocular or periocular infections
14. Active or suspected intraocular inflammation
15. Further clinical contraindications to IMP application (exclusion will be based upon investigator's judgment)
16. Current or previous (within 30 days of enrollment) treatment with another IMP, or participation and/or under follow-up in another clinical trial
17. Previous participation in this clinical trial (except screening failure due to inclusion criterion 2 and/or exclusion criterion 1 and/or 2 and/or 3 and/or 6)
18. Known abuse of alcohol, drugs, or medicinal products
19. Patients unwilling or unable to comply with the requirements of the protocol
20. Lactating women
21. Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment
22. Employees of the sponsor, or employees or relatives of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Response rate at 12 months after IMP application | Month 12
  Response rate at 12 months after IMP application, where response is defined as:
  * no or mild corneal neovascularization (no vessel penetration or vessel penetration up to 1 quadrant, without central cornea) AND
  * no or mild epithelial defects (no corneal erosion or ulcer are present (corneal wounds are closed) or minimal superficial staining)
Assessment of adverse event (AE) occurrence | Up to 24 months.
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Response rate at 3 months after IMP application | Month 3
  Response rate at 3 months after IMP application, where response is defined as:
  * no or mild corneal neovascularization (no vessel penetration or vessel penetration up to 1 quadrant, without central cornea) AND
  * no or mild epithelial defects (no corneal erosion or ulcer are present (corneal wounds are closed) or minimal superficial staining)
Neovascularization | Baseline, week 1, 2, 3, 4, 5, 6, 7, 12, month 6 and 12
  Corneal neovascularization will be assessed as "none" (no blood vessel penetration), "mild" (blood vessel penetration of 1 quadrant, without central cornea involvement), "moderate" (blood vessel penetration of 1 quadrant, with central cornea involvement or blood vessel penetration of 2 or 3 quadrants, with or without central cornea involvement) or "strong" (blood vessel penetration of all quadrants, with or without central cornea involvement).
Epithelial defects | Baseline, week 2, 4, 6, month 3, 6 and 12
  Epithelial defects will be assessed as "none" (no corneal erosion or ulcer are present (corneal wounds are closed)) or "mild" (minimal superficial staining) or "moderate" (dense coalescent staining up to 2 mm in diameter) or "strong" (dense coalescent staining greater than 2 mm in diameter) by means of fluorescein staining.
Ocular symptoms of pain, photophobia, burning | Baseline, week 2, 4, 6, 12, month 6 and 12
  Photophobia and burning will be assessed as "no complaint" (grade 0), "mild" (grade 1), "moderate" (grade 2) or "severe" (grade 3).
  Pain assessment will be done by the patient using a 11-point numerical rating scale ranging between no pain (zero) and worst imaginable pain (ten).
Ocular inflammation | Baseline, week 2, 4, 6, 12, month 6 and 12
  The assessment of inflammation will be categorized as present (yes) or nonexistent (no).
Corneal opacity | Baseline, week 2, 4, 6, 12, month 6 and 12
  Corneal opacification will be assessed as "none" (no corneal opacification), "mild" (corneal opacification in up to 1 quadrant, without central cornea involvement), "moderate" (corneal opacification in 1 quadrant, with central cornea involvement or corneal opacification in 2 or 3 quadrants, with or without central cornea involvement) or "strong" (corneal opacification in all quadrants, with or without central cornea involvement).
  Additional densitometric Pentacam® measurements are optional. Opacity values of the following ring-shaped corneal segments will be record:
  * 0 - 2 mm, 2 - 6 mm, 6 - 10 mm, 10 - 12 mm (anterior, central and posterior corneal layer for each segment)
  * 0 - 2 mm, 2 - 6 mm, 6 - 10 mm, 10 - 12 mm (full thickness average for each segment)
  * Anterior layer of the complete cornea (0 - 12 mm)
  * Central layer of the complete cornea (0 - 12 mm)
  * Posterior of the complete cornea (0 - 12 mm)
  * Overall cornea (0 - 12 mm, full thickness)
Visual acuity | Baseline, week 2, 4, 6, 12, month 6 and 12
  Clarity of vision.
Quality of life assessment | Baseline, week 12, month 12
  Quality of life (visual function questionnaire-25 [VFQ-25]) questionnaire to be answered.
Physical examination | Baseline, week 12, month 12
  A full physical examination will be performed at week 12 and abnormal physical examination results will be evaluated and reported as AEs.
Tonometry | Baseline,week 1, 3, 7 and 12
Vital signs: Body temperature at Baseline, week 12, month 12 | Baseline, week 12, month 12
  Body temperature at Baseline, week 12 and month 12 will be evaluated.
Vital signs: Blood pressure at Baseline, week 12, month 12 | Baseline, week 12, month 12
  Blood pressure at Baseline, week 12 and month 12 will be evaluated.
Vital signs: Heart rate at Baseline, week 12, month 12 | Baseline, week 12, month 12
  Heart rate at Baseline, week 12 and month 12 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd U. Auffarth, Prof.Dr.med., Principal Investigator — Universitäts-Klinikum Heidelberg, Kopfklinik, Heidelberg, Germany
Locations (5):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States
- Germany (4):
  - Universitäts-Klinikum Köln, Augenklinik, Cologne
  - Universitäts-Klinikum Heidelberg, Kopfklinik, Heidelberg
  - Universitäts-Klinikum Jena, Augenklinik, Jena
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Augenklinik und Poliklinik, Mainz

IPD SHARING:
Plan to Share IPD: No